CLINICAL TRIAL: NCT02586688
Title: A Randomized, Sham-Controlled Trial Evaluating the Safety and Effectiveness of NeuroStar® Transcranial Magnetic Stimulation (TMS) Therapy in Depressed Adolescents
Brief Title: Safety and Effectiveness of NeuroStar® Transcranial Magnetic Stimulation (TMS) Therapy in Depressed Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 44-02219-000
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: child depression; depression; Transcranial Magnetic Stimulation; Adolescent Major Depressive Disorder; TMS; adolescent depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I TMS Active (Active Comparator): Blinded Active TMS coil (Phase I). Active NeuroStar® Transcranial Magnetic Stimulation (TMS)
  Interventions: Device: Active NeuroStar® Transcranial Magnetic Stimulation (TMS)
- Phase I TMS Sham (Sham Comparator): Blinded Sham TMS coil (Phase I) Sham NeuroStar® Transcranial Magnetic Stimulation (TMS)
  Interventions: Device: Sham NeuroStar® Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Active NeuroStar® Transcranial Magnetic Stimulation (TMS) — Compare active NeuroStar® coil with sham NeuroStar® coil.
  Other Names: TMS; NeuroStar®
  Arms: Phase I TMS Active
Device: Sham NeuroStar® Transcranial Magnetic Stimulation (TMS) — Compare active NeuroStar® coil with sham NeuroStar® coil.
  Other Names: TMS; NeuroStar®
  Arms: Phase I TMS Sham

SUMMARY:
To evaluate the safety and efficacy of daily, active Neurostar® TMS (when compared with sham treatment) in adolescents meeting criteria for Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
To evaluate the antidepressant effects of daily, active TMS (when compared with sham treatment) in adolescents meeting criteria for Major Depressive Disorder, single or recurrent episode.

Secondary:

To evaluate the acute and long term safety of TMS treatment in adolescent MDD subjects.

To evaluate the durability of benefit of TMS treatment over the course of 6 months in subjects who received clinical benefit from acute treatment course(s) .

To evaluate the benefit of daily, active, open-label TMS in Phase I subjects who did not receive protocol-defined clinical benefit; as new acute treatment (sham to active) or as extended treatment course (blinded active to open label active) .

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of unipolar major depressive disorder, in a current major depressive episode, without psychotic features
* Duration of current episode of depression ≥4 weeks and ≤3 years
* Clinical Global Impression - Severity of Illness ≥ 4
* Resistance to antidepressant treatment in a discrete illness episode
* HAMD24 Item 1 ≥ 2 and total score ≥ 20
* Subjects able to commit to protocol visit schedule
* At the end of the baseline visit, subject must have a HAMD24 score of ≥ 18 and change in score may not be ≥ 25% decrease from that seen at the screening visit

Exclusion Criteria:

* Prior TMS, vagus nerve stimulation (VNS), or electroconvulsive therapy (ECT)
* Contraindication to TMS
* Cardiac pacemakers, implanted medication pumps, intracardiac lines
* History of neurological disorder
* Unstable medical conditions
* Any psychiatric disorder, which in the judgement of the Investigator may hinder the subject in completing the procedures required by the study protocol.
* Significant acute suicide risk
* Inability to locate and quantify a motor threshold
* If sexually active female, not on an accepted method of birth control.
* Diagnoses of the following conditions (current unless otherwise stated):

  * Depression secondary to a general medical condition, or substance induced:
  * Seasonal pattern of depression as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
  * Any psychotic disorder (lifetime), including history of schizophrenia, schizoaffective disorder, other psychosis, psychotic features in this or previous episodes, amnestic disorder,
  * Intellectually disabled,
  * Substance dependence or abuse within the past year (except nicotine or caffeine),
  * Bipolar disorder,
  * Obsessive compulsive disorder (lifetime),
  * Post-traumatic stress disorder (lifetime),
  * Eating disorder (lifetime).

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2015-10; Primary Completion 2018-01 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Croarkin, MD, Principal Investigator — Mayo Clinic; Karen Heart, Study Director — Neuronetics
Locations (13):
- United States (13):
  - Dothan Behavioral Medicine, Dothan, Alabama
  - UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Rocky Mountain TMS, Grand Junction, Colorado
  - Florida Clinical Practice Association, Inc., Gainesville, Florida
  - Anchor Neuroscience, Pensacola, Florida
  - Beacon Medical Group, South Bend, Indiana
  - Integrative Psychiatry, Louisville, Kentucky
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Result] Carpenter LL, Janicak PG, Aaronson ST, Boyadjis T, Brock DG, Cook IA, Dunner DL, Lanocha K, Solvason HB, Demitrack MA. Transcranial magnetic stimulation (TMS) for major depression: a multisite, naturalistic, observational study of acute treatment outcomes in clinical practice. Depress Anxiety. 2012 Jul;29(7):587-96. doi: 10.1002/da.21969. Epub 2012 Jun 11. PMID 22689344
- [Result] Wall CA, Croarkin PE, Sim LA, Husain MM, Janicak PG, Kozel FA, Emslie GJ, Dowd SM, Sampson SM. Adjunctive use of repetitive transcranial magnetic stimulation in depressed adolescents: a prospective, open pilot study. J Clin Psychiatry. 2011 Sep;72(9):1263-9. doi: 10.4088/JCP.11m07003. PMID 21951987

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data regarding Phase 2 and phase 3 of the study is not available. Primary analyses for the phase 1 data showed the study didnt meet its primary end point and hence no further analyses was done.
Groups:
- TMS Active: Blinded Active TMS coil (Phase I). Active NeuroStar® Transcranial Magnetic Stimulation (TMS)
  Active NeuroStar® Transcranial Magnetic Stimulation (TMS): Compare active NeuroStar® coil with sham NeuroStar® coil.
- TMS Sham: Blinded Sham TMS coil (Phase I) Sham NeuroStar® Transcranial Magnetic Stimulation (TMS)
  Sham NeuroStar® Transcranial Magnetic Stimulation (TMS): Compare active NeuroStar® coil with sham NeuroStar® coil.
Period: Overall Study
Arm/Group | TMS Active | TMS Sham
Started | 54 | 58
Completed | 48 | 55
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- TMS Active Arm: Blinded Active TMS coil Active NeuroStar® Transcranial Magnetic Stimulation (TMS)
  Active NeuroStar® Transcranial Magnetic Stimulation (TMS): Compare active NeuroStar® coil with sham NeuroStar® coil.
- TMS Sham Arm: Blinded Sham TMS coil Sham NeuroStar® Transcranial Magnetic Stimulation (TMS)
  Sham NeuroStar® Transcranial Magnetic Stimulation (TMS): Compare active NeuroStar® coil with sham NeuroStar® coil.
- Total: Total of all reporting groups
Arm/Group | TMS Active Arm | TMS Sham Arm | Total
Number analyzed (Participants) | 48 | 55 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 35 | 62
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — In total, 103 patients met criteria for modified intent to treat (mITT) of at least 1 treatment and a posttreatment HAM-D-24 rating.
  Although these patients did not meet inclusion criteria, they were included in the analyses given the importance of the safety data and following the modified intent-to-treatment principal as pre-specified for the efficacy analysis
  years | 17.6 (2.28) | 17.2 (2.22) | 17.4 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 67
  Male | 18 | 18 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 48 | 55 | 103
The Hamilton Rating Scale for Depression (HRSD) [Mean (Standard Deviation); unit: units on a scale] — HAM-D-24 or 24-item Hamilton Depression Rating Scale; Total score rage is 0-76 and Lower score is better
  units on a scale | 28.8 (5.75) | 29.5 (6.69) | 29.15 (6.22)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale-24(HAMD24) Total Score Change From Baseline Value.
Description: The Hamilton Rating Scale for Depression (HRSD), also called the Hamilton Depression Rating Scale (HDRS), sometimes also abbreviated as HAM-D, is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.HAM-D-24 24-item Hamilton Depression Rating Scale; Lower score is better (76 to 0)
Time Frame: 6 weeks
Population: Open Label population not analyzed for primary treatment effect. Continued treatment for maintenance
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase I TMS Active | Phase I TMS Sham
Number analyzed (Participants) | 48 | 55
score on a scale | -11.1 (2.03) | -10.6 (2.00)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Summary of AEs during the first 6 weeks post randomization to active TMS vs Sham
Groups:
- TMS Active Arm: Blinded Active TMS coil . Active NeuroStar® Transcranial Magnetic Stimulation (TMS)
  Active NeuroStar® Transcranial Magnetic Stimulation (TMS): Compare active NeuroStar® coil with sham NeuroStar® coil.
Arm/Group | TMS Active Arm | TMS Sham Arm
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/58
Serious Adverse Events (participants affected / at risk) | 3/54 | 1/58
Other Adverse Events (participants affected / at risk) | 31/54 | 19/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Active Arm (N=54) | TMS Sham Arm (N=58)
Suicide Attempt (classified as definitely not related to the study device) (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation- not related to study device (Psychiatric disorders) | 1 (1) | 1 (1)
Worsening Depression- classified as definitely not related to the study device (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Active Arm (N=54) | TMS Sham Arm (N=58)
Eye Pain (Eye disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (3) — Nausea and Vomiting
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Twitching Facial (Gastrointestinal disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 17 (17) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT02586688/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT02586688/SAP_001.pdf